CLINICAL TRIAL: NCT04234997
Title: Suvorexant to Reduce Symptoms of Nicotine Use: A Double-blind, Placebo-controlled Study
Brief Title: Suvorexant to Reduce Symptoms of Nicotine Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Robert Suchting, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-19-0966
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suvorexant 20 mg (Experimental)
  Interventions: Drug: Suvorexant 20 mg
- Suvorexant 0mg (Placebo Comparator)
  Interventions: Drug: Suvorexant 0mg

INTERVENTIONS:
Drug: Suvorexant 20 mg — Participants will be advised to take the medication at 10PM for 7 days.Participants will be instructed to stop smoking by 10 pm the day before, in order to ensure they meet the breath CO criterion (CO ≤ 4 ppm) indicating overnight abstinence.
  Arms: Suvorexant 20 mg
Drug: Suvorexant 0mg — Participants will be advised to take the medication at 10PM for 7 days.Participants will be instructed to stop smoking by 10 pm the day before, in order to ensure they meet the breath CO criterion (CO ≤ 4 ppm) indicating overnight abstinence.
  Arms: Suvorexant 0mg

SUMMARY:
The purpose of this study is to assess the impact of suvorexant on established measures of smoking relapse risk (craving,withdrawal, stress reactivity, latency to self-administration) and to validate the somnolent effect of suvorexant on sleep metrics in a sample of individuals with tobacco use disorder

ELIGIBILITY:
Inclusion Criteria:

* non-treatment seeking cigarette smokers that report smoking atleast 10 cigarettes per day

Exclusion Criteria:

* greater than mild substance use disorder on drugs other than nicotine
* a Diagnostic and Statistical Manual of Mental Disorders(DSM)-IV axis I psychiatric disorder or neurological disease or disorder requiring ongoing treatment and/or making study participation unsafe
* significant current suicidal or homicidal ideation - medical conditions contraindicating administration of suvorexant (e.g., severe pulmonary disease, severe cardiovascular disease or clinically abnormal EEG, severe liver or kidney disease, seizure disorder, or sleep disorder - particularly narcolepsy)
* taking medications known to have significant drug interactions with the study medication(s) (e.g., Monoamine oxidase inhibitors(MAO) inhibitors, anticonvulsants, haloperidol, phenothiazines, anesthetics, and all sedatives)
* currently or recently (last 3 months) treated for substance use [other than nicotine] or another psychiatric condition
* conditions of probation or parole requiring reports of drug use to officers of the court
* impending incarceration
* pregnant or nursing for female patients
* inability to read, write, or speak English [required for lab tasks and psychometric scales]
* unwillingness to sign a written informed consent form
* subjects with alcohol use disorders or report recent problem drinking (5/4 drinks for males/females in < 2.5 hours or > 10 alcoholic drinks per week)
* any illness,condition, or use of medications which in the opinion of the PI and/or admitting physician would preclude safe and/or successful completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Suchting, Ph.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 14 enrolled participants, 11 were randomized and 3 withdrew from the study before randomization.
Period: Overall Study
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Started | 5 | 6
Completed | 3 | 5
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: include all who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.60 (7.92) | 46.67 (7.15) | 49.36 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 3 | 4 | 7
  White | 2 | 1 | 3
  Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11
Years of Education [Mean (Standard Deviation); unit: years] | 12.20 (0.45) | 12.83 (1.83) | 12.55 (1.37)
Nicotine dependence as assessed by the Fagerstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: score on a scale] — The Fagerström Test for Nicotine Dependence (FTND) is a standard instrument used to assess the intensity of physical addiction to nicotine. Total scores range from 0 to 10, with higher scores indicating greater nicotine dependence.
  score on a scale | 5.80 (1.64) | 6.17 (1.94) | 6.00 (1.73)
Cognitive ability as assessed by Shipley 2- Composite B [Mean (Standard Deviation); unit: score on a scale] — The Shipley 2- Composite B measures cognitive ability. The total score ranges from 25 to 145, higher score indicating higher cognitive ability.
  score on a scale | 91.00 (14.07) | 98.00 (10.83) | 94.82 (12.29)

OUTCOME MEASURES:

1. Primary Outcome: Stress as Assessed by a Visual Analog Scale (VAS) for Stress
Description: The VAS total score ranges from 1(none) to 10(extreme stress);a higher score indicating a worse outcome.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
score on a scale | 3.4 (2.07) | 3 (2.61)

2. Primary Outcome: Stress as Assessed by a Visual Analog Scale (VAS) for Stress
Description: The VAS total score ranges from 1(none) to 10(extreme stress);a higher score indicating a worse outcome.
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
score on a scale | 3.33 (2.89) | 3.2 (2.39)

3. Primary Outcome: Change in Stress Reactivity as Assessed by Heart Rate During the Cold Pressor Test (CPT)
Description: During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. Heart rate will be collected pre CPT (about 15 minutes before cold pressor task) and post CPT (about 2 minutes after the start of the cold pressor task). The change in Heart rate will be reported as [(Heart rate post cold pressor task) - (Heart rate pre cold pressor task)].
Time Frame: Day 1 baseline (about 15 minutes before cold pressor task) and about 2 minutes after the start of the cold pressor task
Measure: Mean (Standard Deviation); unit: beats per minutes (bpm)
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
beats per minutes (bpm) | 5 (1.581) | 9.5 (3.728)

4. Primary Outcome: Change in Stress Reactivity as Assessed by Heart Rate During the Cold Pressor Test (CPT)
Description: as for outcome 3
Time Frame: Day 8 baseline (about 15 minutes before cold pressor task) and about 2 minutes after the start of the cold pressor task
Measure: Mean (Standard Deviation); unit: beats per minutes (bpm)
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
beats per minutes (bpm) | 3.667 (1.528) | 9 (4.183)

5. Primary Outcome: Change in Stress Reactivity as Assessed by Cortisol During the Cold Pressor Test (CPT)
Description: During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. Saliva samples will be collected pre CPT (about 15 minutes before cold pressor task) and post CPT (about 30 minutes after the start of the cold pressor task), and cortisol levels in the saliva samples will be assessed. The change in cortisol level will be reported as [(cortisol level at post cold pressor task) - (cortisol level pre cold pressor task)].
Time Frame: Day 1 baseline (about 15 minutes before cold pressor task) and about 30 minutes after the start of the cold pressor task, Day 8 baseline (about 15 minutes before cold pressor task) and about 30 minutes after the start of the cold pressor task
Population: All cortisol samples were compromised during collection and storage due to cross-contamination between control and experimental samples. As a result, the samples could not be processed, and no outcome data were collected.
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Smoking as Assessed by Latency to Self-Administration During the Smoking Relapse Assessment
Description: Latency to self-administration is defined as the time (in minutes) from the beginning of the relapse assessment session until the participant initiates smoking their first cigarette.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
minutes | 56.8 (4.44) | 22.67 (22.99)

7. Primary Outcome: Smoking as Assessed by Number of Self-Administrated Cigarettes During the Smoking Relapse Assessment
Description: The outcome measure is the number of cigarettes self-administered by each participant during the Smoking Relapse Assessment.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
cigarettes | 0.8 (1.3) | 1.33 (0.52)

8. Primary Outcome: Change in Sleep Quality as Assessed by the Garmin Vivosmart3 Actigraphy Device
Description: Quality defined as proportion of time in deep sleep. Change in sleep quality is reported as [(Day 8 Sleep Quality ) - (Day 1 Sleep quality)]
Time Frame: Day 1, Day 8
Population: Data were not collected from 3 participants in the Suvorexant 20 mg arm and Data were not collected for 5 participants in the Suvorexant 0mg due to device malfunction and/or user error.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 2 | 1
minutes | -0.038 (0.1) | 0.4

9. Primary Outcome: Change in Sleep Duration as Assessed by the Garmin Vivosmart3 Actigraphy Device
Description: Duration as the total amount of time asleep. Change in sleep duration is reported as [(Day 8 Sleep Duration ) - (Day 1 Sleep Duration)]
Time Frame: Day 1, Day 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 2 | 1
minutes | -195.5 (229.8) | 79

10. Primary Outcome: Change in Sleep Restlessness as Assessed by the Garmin Vivosmart3 Actigraphy Device
Description: Restlessness as the number of times waking up during sleep. Change in sleep restlessness is reported as [(Day 8 Sleep restlessness) - (Day 1 Sleep restlessness]
Time Frame: Day 1, Day 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: number of times awake
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 2 | 1
number of times awake | 0.5 (0.707) | 7

11. Primary Outcome: Smoking as Assessed by Number of Self-Administrated Cigarettes During the Smoking Relapse Assessment
Description: as for outcome 7
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: cigarettes
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
cigarettes | 1.33 (2.31) | 1.4 (0.55)

12. Primary Outcome: Smoking as Assessed by Latency to Self-Administration During the Smoking Relapse Assessment
Description: as for outcome 6
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
minutes | 56.67 (5.77) | 16.2 (22.02)

13. Primary Outcome: Nicotine Craving as Assessed by the Questionnaire of Smoking Urgers (QSU-brief)
Description: The Questionnaire of Smoking Urgers (QSU-brief) total score ranges from 10 to 70, higher score indicates greater nicotine craving.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
score on a scale | 45.8 (12.24) | 36.67 (14.92)

14. Primary Outcome: Nicotine Craving as Assessed by the Questionnaire of Smoking Urgers (QSU-brief)
Description: as for outcome 13
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
score on a scale | 47.67 (17.21) | 39.8 (11.17)

15. Secondary Outcome: Stress as Assessed by the Depression-Anxiety-Stress 21 (DASS21) Self-Report Questionnaire - Stress Subscale
Description: The Stress Subscale of the Depression, Anxiety and Stress scale (DASS-21) assesses stress levels. Total score on the DASS-21 stress subscale ranges from 0 to 21, with a higher score indicating higher stress.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
score on a scale | 0.8 (0.84) | 3.5 (2.74)

16. Secondary Outcome: Stress as Assessed by the Depression-Anxiety-Stress 21 (DASS21) Self-Report Questionnaire - Stress Subscale
Description: as for outcome 15
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
score on a scale | 1.33 (1.15) | 5.2 (4.15)

17. Secondary Outcome: Stress as Assessed by the Personal Stress Scale (PSS)
Description: The Personal Stress Scale (PSS) total score ranges from 0 to 40, a higher score indicating greater stress.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
score on a scale | 17.2 (4.15) | 19 (2.61)

18. Secondary Outcome: Stress as Assessed by the Personal Stress Scale (PSS)
Description: The Personal Stress Scale (PSS) total score ranges from 0 to 40, a higher score indicating greater stress.
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
score on a scale | 18 (6.24) | 17.4 (2.88)

19. Secondary Outcome: Change in Stress Reactivity as Assessed by Systolic Blood Pressure During the Cold Pressor Test (CPT)
Description: During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. Systolic Blood Pressure will be collected pre CPT (about 15 minutes before cold pressor task) and post CPT (about 2 minutes after the start of the cold pressor task). The change in Systolic Blood Pressure will be reported as [( Systolic Blood Pressure at post cold pressor task) - (Systolic Blood Pressure at pre cold pressor task)].
Time Frame: Day 1 baseline (about 15 minutes before cold pressor task) and about 2 minutes after the start of the cold pressor task
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
millimeters of mercury (mmHg) | 17.6 (18.94) | 27.833 (10.572)

20. Secondary Outcome: Change in Stress Reactivity as Assessed by Systolic Blood Pressure During the Cold Pressor Test (CPT)
Description: During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. Systolic Blood Pressure will be collected pre CPT (about 15 minutes before cold pressor task) and post CPT (about 2 minutes after the start of the cold pressor task) The change in Systolic Blood Pressure will be reported as [( Systolic Blood Pressure at post cold pressor task) - (Systolic Blood Pressure at pre cold pressor task)].
Time Frame: Day 8 baseline (about 15 minutes before cold pressor task) and about 2 minutes after the start of the cold pressor task
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
millimeters of mercury (mmHg) | 18 (11.358) | 16 (8.276)

21. Secondary Outcome: Change in Stress Reactivity as Assessed by Diastolic Blood Pressure During the Cold Pressor Test (CPT)
Description: During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. Diastolic Blood Pressure will be collected pre CPT (about 15 minutes before cold pressor task) and post CPT (about 2 minutes after the start of the cold pressor task). The change in Diastolic Blood Pressure will be reported as [( Diastolic Blood Pressure at post cold pressor task) - (Diastolic Blood Pressure at pre cold pressor task)].
Time Frame: Day 1 baseline (about 15 minutes before cold pressor task) and about 2 minutes after the start of the cold pressor task
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
millimeters of mercury (mmHg) | 7.4 (9.449) | 22.667 (8.165)

22. Secondary Outcome: Change in Stress Reactivity as Assessed by Diastolic Blood Pressure During the Cold Pressor Test (CPT)
Description: During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. Diastolic Blood Pressure will be collected pre CPT (about 15 minutes before cold pressor task) and post CPT (about 2 minutes after the start of the cold pressor task).The change in Diastolic Blood Pressure will be reported as [( Diastolic Blood Pressure at post cold pressor task) - (Diastolic Blood Pressure at pre cold pressor task)].
Time Frame: Day 8 baseline (about 15 minutes before cold pressor task) and about 2 minutes after the start of the cold pressor task
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
millimeters of mercury (mmHg) | 9.667 (3.512) | 14.8 (4.382)

23. Secondary Outcome: Sleep Quality as Assessed by the Patient-Reported Outcomes Measurement Information System(PROMIS) Sleep Disturbance Short Form
Description: Patient-Reported Outcomes Measurement Information System(PROMIS) Sleep Disturbance Short Form total score ranges from 8 to 40, a higher score indicating worse sleep quality.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
score on a scale | 16.4 (6.07) | 18.83 (8.89)

24. Secondary Outcome: Sleep Quality as Assessed by the Patient-Reported Outcomes Measurement Information System(PROMIS) Sleep Disturbance Short Form
Description: as for outcome 23
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
score on a scale | 16 (5.2) | 21.4 (10.76)

25. Secondary Outcome: Sleep Quality as Assessed by the Epworth Sleepiness Scale (ESS)
Description: The Epworth Sleepiness Scale (ESS) total score ranges from 0 to 24, a higher score indicating worse sleep quality.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
score on a scale | 9.8 (6.61) | 7.67 (5.35)

26. Secondary Outcome: Sleep Quality as Assessed by the Epworth Sleepiness Scale (ESS)
Description: The Epworth Sleepiness Scale (ESS) total score ranges from 0 to 24, a higher score indicating worse sleep quality.
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
score on a scale | 12.67 (8.62) | 11 (6.04)

27. Secondary Outcome: Withdrawal Severity as Assessed by the Minnesota Nicotine Withdrawal Questionnaire (MNWQ)
Description: The Minnesota Nicotine Withdrawal Questionnaire (MNWQ) total score ranges from 0 to 36 with higher scores indicating greater withdrawal symptoms.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
score on a scale | 9.6 (7.8) | 6.67 (3.93)

28. Secondary Outcome: Withdrawal Severity as Assessed by the Minnesota Nicotine Withdrawal Questionnaire (MNWQ)
Description: as for outcome 27
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
score on a scale | 7 (5.29) | 11.6 (7.02)

29. Secondary Outcome: Anxiety a Measured by the Hamilton Anxiety Rating Scale (HAM-A)
Description: The Hamilton Anxiety Rating Scale (HAM-A) total score ranges from 0 to 56, a higher score indicating greater anxiety.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
score on a scale | 2.8 (2.05) | 3.17 (1.47)

30. Secondary Outcome: Anxiety a Measured by the Hamilton Anxiety Rating Scale (HAM-A)
Description: The Hamilton Anxiety Rating Scale (HAM-A) total score ranges from 0 to 56, a higher score indicating greater anxiety.
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
score on a scale | 2.33 (3.21) | 3 (1.22)

31. Secondary Outcome: Sleep Quality as Assessed by the Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) total score ranges from 0 to 21, a higher score indicates worse sleep quality.
Time Frame: Day 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
score on a scale | 8 (2.55) | 8.67 (5.54)

32. Secondary Outcome: Sleep Quality as Assessed by the Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) total score ranges from 0 to 21, a higher score indicates worse sleep quality.
Time Frame: Day 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
score on a scale | 7 (2) | 9.8 (4.44)

33. Secondary Outcome: Anxiety as Assessed by the Depression-Anxiety-Stress 21 (DASS21) Self-Report Questionnaire - Anxiety Subscale
Description: The Anxiety Subscale of the Depression, Anxiety and Stress scale (DASS-21) assesses anxiety levels. Total score on the DASS-21 stress subscale ranges from 0 to 21, with a higher score indicating greater anxiety.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
score on a scale | 0.8 (1.3) | 2.5 (2.17)

34. Secondary Outcome: Anxiety as Assessed by the Depression-Anxiety-Stress 21 (DASS21) Self-Report Questionnaire - Anxiety Subscale
Description: as for outcome 33
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
score on a scale | 0.67 (0.58) | 3 (3)

35. Secondary Outcome: Change in Stress as Assessed by Visual Analog Scale (VAS) for Stress During the Cold Pressor Test (CPT)
Description: During the cold pressor task (CPT), participants will submerge their dominant arm in an ice-water bath for up to 2 minutes. The VAS total score ranges from 1(none) to 10(extreme stress);a higher score indicating a worse outcome. Visual Analog Scale (VAS) for stress score will be collected before and after the CPT. The change in Stress will be reported as [( Visual Analog Scale (VAS) for stress score at post cold pressor task) - (Visual Analog Scale (VAS) for stress score at pre cold pressor task)].
Time Frame: Day 1 baseline (about 15 minutes before cold pressor task) and about 30 minutes after the start of the cold pressor task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 5 | 6
score on a scale | 0 (0.707) | 0 (0)

36. Secondary Outcome: Change in Stress as Assessed by Visual Analog Scale (VAS) for Stress During the Cold Pressor Test (CPT)
Description: as for outcome 35
Time Frame: Day 8 baseline (about 15 minutes before cold pressor task) and about 30 minutes after the start of the cold pressor task
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
Number analyzed (Participants) | 3 | 5
score on a scale | 1 (1) | -0.2 (0.447)

ADVERSE EVENTS:
Time Frame: Up to 8 Days
Arm/Group | Suvorexant 20 mg | Suvorexant 0mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT04234997/Prot_SAP_000.pdf